CLINICAL TRIAL: NCT06697171
Title: The Comparative Effectiveness of Different Conflict-of-interest Disclosures Displayed on Social Media Posts by Registered Dietitians on Public Transparency, Trust and Purchasing Intentions: A Randomized Controlled Experiment
Brief Title: Effectiveness of Conflict-of-interest Disclosures on Trust, Credibility and Transparency When Displayed on Social Media Posts From Registered Dietitians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ontario Institute of Technology (Other)
Responsible Party: Principal Investigator, JoAnne Arcand, Principal Investigator, University of Ontario Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17546
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Registered Dietitian; Conflict of Interest; Trust; Credibility; Transparency
Keywords: Registered Dietitian; Conflict of Interest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (Active Comparator): No COI Disclosure (Control). Only @brandname is tagged in the social media post narrative body.
  Interventions: Other: Control
- Group 1 Not an Ad Disclosure (Experimental): Disclosure includes @brandname and #NotAnAd in the social media post narrative body.
  Interventions: Other: Group 1 Not an ad disclosure
- Group 2 Basic Disclosure (Experimental): Disclosure includes @brandname and #ad in the narrative body of the social media post.
  Interventions: Other: Group 2 Basic Disclosure
- Group 3 Basic + Paid Partnership Disclosure (Experimental): Disclosure includes a branded "paid partnership" in the header and a tag for the industry partner, @brandname and #ad immediately at the beginning of the post, and #ad and #sponsored at the bottom of the narrative body of the social media post.
  Interventions: Other: Group 3 Basic + Paid Partnership Disclosure
- Group 4 Basic + Paid Partnership + Image label (Experimental): Disclosure includes the same attributes as Group 3, with the addition of #ad appearing on the post image itself.
  Interventions: Other: Group 4 Basic + Paid Partnership + Image label

INTERVENTIONS:
Other: Group 1 Not an ad disclosure — Same social media post viewed as all other groups. @brandname in the narrative body of the social media post; #NotAnAd in the narrative body of the social media post
  Arms: Group 1 Not an Ad Disclosure
Other: Group 2 Basic Disclosure — Same social media post viewed as all other groups. @brandname in the narrative body of the social media post; #ad in the narrative body of the social media post
  Arms: Group 2 Basic Disclosure
Other: Group 3 Basic + Paid Partnership Disclosure — Same social media post viewed as all other groups. COI disclosures include "paid partnership" in the header and a tag for the industry partner; @brandname and #ad immediately at the beginning of the narrative body of the social media post;
  #ad and #sponsored at the bottom of the narrative body of the social media post.
  Arms: Group 3 Basic + Paid Partnership Disclosure
Other: Control — No COI disclosure elements (i.e. no hashtags ). Only the @brandname is included within the narrative body of the social media post.
  Arms: Control
Other: Group 4 Basic + Paid Partnership + Image label — Same social media post viewed as all other groups. COI disclosures include "paid partnership" in the header and a tag for the industry partner; @brandname and #ad immediately at the beginning of the narrative body of the social media post; #ad and #sponsored at the bottom of the narrative body of the social media post; #ad (black text, white background) appears on the photo associated with the social media post
  Arms: Group 4 Basic + Paid Partnership + Image label

SUMMARY:
There is limited research to inform policies and guidelines related to disclosing conflicts of interest on social media by healthcare professionals, including Registered Dietitians (RDs). This trial investigates mock social media posts by an RD to examine the impact of varying forms of conflict-of-interest (COI) disclosures. The disclosures tested are based on the Canadian Ad Standards "Influencer Marketing Disclosure Guidelines" and are incorporated into recommendations established by the provincial dietetic regulatory bodies for RDs. Specific outcomes evaluated include the public's ability to identify a COI; trust in the RD; credibility of the RD; transparency of the social media post and; purchasing and consumption intentions of the product endorsed by an RD in the post.

DETAILED DESCRIPTION:
This study is a randomized controlled experiment embedded within an online cross-sectional survey entitled the Canadian Nutrition and Health Survey (CNHS). A sample of 3,380 Canadian adults from all Canadian provinces (ages ≥18 years, who own a computer, and have an email address) will be recruited by Leger Marketing Inc. as part of the CNHS. Participants will be randomized to one of five experimental groups that include a mock social media post with different variations of COI reporting, based on the Ad Standards (of Canada) Influencer Marketing Disclosure Guidelines. Each participant will be randomized to view one version (group) of the mock Instagram post, all of which feature the same RD promoting the nutritional benefits of a mock soy milk product. Participants will also have the opportunity to view the RD's Instagram account profile, which is consistent across all experimental groups. All participants will have as much time as needed to view the post and account profile.

As stated previously, the experimental groups vary by the extent to which the conflict of interest is reported (see below):

* Group 1 Not an ad disclosure: COI disclosure includes @brandname and #NotAnAd in the narrative body of the social media post.
* Group 2 Basic Disclosure: COI disclosure includes @brandname and #ad in the narrative body of the social media post.
* Group 3 Basic + Paid Partnership Disclosure: COI disclosure accompanied by a branded "paid partnership" in the header and a tag for the industry partner, @brandname and #ad immediately at the beginning of the post, and #ad and #sponsored at the bottom of the narrative body of the social media post.
* Group 4 Basic + Paid Partnership + Image label: COI disclosure includes the same characteristics as Group 3, with the addition of #ad appearing on the post image itself.
* Group 5 Control group: is a control with no COI disclosure elements (i.e. no hashtags and only the @brandname included within the narrative body of the social media post).

The primary outcome is the ability of a participant to identify if COI disclosures exist within the social media post. The secondary outcomes include participants' trust in the RD in the social media post, credibility of the RD in the social media post, participants' buying and consumption intentions, and transparency of COI reporting by the RD. Tertiary outcomes include the participants' recommendation of the food item endorsed by the RD to others, participants' engagement with the social media post, and participants' view of the healthfulness of a product endorsed by the RD.

It is hypothesized that, compared to the control condition, participants will rate all experimental conditions as having a conflict of interest. The experimental conditions will be rated more transparent and trustworthy, with the RD in the social media post being rated as more credible, and with greater purchasing/consumption intentions.

ELIGIBILITY:
Inclusion Criteria:

Participants are included if:

* are ≥18 years
* own a computer,
* have an email address
* speak/write in English/French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3409 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Conflict of Interest | Measured after 5-10 minutes of exposure to the social media post
  Participant identification of COI will be:
  * Assessed by the statement "I believe the person in the post has a conflict of interest"
  * Evaluated on a 5-point Likert Scale from Strongly Disagree (1) to Strongly Agree (5). There is no "not applicable" option.

SECONDARY OUTCOMES:
Trust | Measured after 5-10 minutes of exposure to the social media post
  •Trust of the RDs post will be:
  * Assessed by the statements "I trust the person in this post" and "I believe the post is true". This is also assessed using an open-ended question.
  * Evaluated on a 5-point Likert Scale from Strongly Disagree (1) to Strongly Agree (5). There is no "not applicable" option.
Credibility | Measured after 5-10 minutes of exposure to the social media post
  • The RD's credibility will be:
  * Assessed by the statement "The person in this post is qualified to provide this information".
  * Evaluated on a 5-point Likert Scale from Strongly Disagree (1) to Strongly Agree (5). There is no "not applicable" option.
Purchasing Intentions | Measured after 5-10 minutes of exposure to the social media post
  • The participants' purchasing intentions of a product after viewing the post will be:
  * Assessed by the statement: How likely you would "Buy the food item in the post" and "I am more likely to buy a product if a Registered Dietitian has endorsed it" (both will be reviewed separately)
  * Evaluated on a 5-point Likert Scale from Very Unlikely (1) to Very Likely (5). There is no "not applicable" option.
Consumption Intentions | Measured after 5-10 minutes of exposure to the social media post
  • The participants' consumption intentions of a product after seeing the RDs post will be:
  * Assessed by the statement: How likely you would "Consume the food item in the post"
  * Evaluated on a 5-point Likert Scale from Very Unlikely (1) to Very Likely (5). There is no "not applicable" option.
Transparency | Measured after 5-10 minutes of exposure to the social media post
  • Transparency of the RDs post will be:
  * Assessed by the statement "The food item is being endorsed"
  * Evaluated on a 5-point Likert Scale from Strongly Disagree (1) to Strongly Agree (5). There is no "not applicable" option.

OTHER OUTCOMES:
Recommendation | Measured after 5-10 minutes of exposure to the social media post
  • Participants' recommendation a product endorsed by an RD will be:
  * Assessed by the statement "Recommend the food item in the post to others (e.g., family, friends)"
  * Evaluated on a 5-point Likert Scale from Very Unlikely (1) to Very Likely (5). There is no "not applicable" option.
Engagement with the post | Measured after 5-10 minutes of exposure to the social media post
  • Participants' engagement with the social media post by an RD:
  * Assessed by the statement, "Like, comment or share this post on social media"
  * Evaluated on a 5-point Likert Scale from Very Unlikely (1) to Very Likely (5). There is no "not applicable" option.
Healthfulness | Measured after 5-10 minutes of exposure to the social media post
  • Participants' view of healthfulness of a product will be:
  * Assessed by the statements, "How healthy do you think soy milk is" and "After reviewing the post, how healthy do you think soy milk is?"
  * Evaluated on a 5-point Likert Scale from Not at all healthy (1) to Very healthy (5). There is no "not applicable" option.
Frequency | Measured after 5-10 minutes of exposure to the social media post
  Frequency of consumption of soy milk was:
  * Assessed by the statement "How often do you have soy milk?"
  * Evaluated on a 5-point Likert Scale from Never (1) to Always (5). There is no "not applicable" option.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ontario Institute of Technology, Oshawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided